CLINICAL TRIAL: NCT04827316
Title: Clinical Utility and Outcome Prediction of Cardiovascular Computed Tomography (PREDICT-CT)
Acronym: PREDICT-CT
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00058
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Coronary Arteriosclerosis; Coronary; Ischemic
Keywords: Cardiovascular Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing clinically indicated CCTA: Patients undergoing clinically indicated CCTA

SUMMARY:
In this study the investigators retrospectively and prospectively collect information from enrolled subjects undergoing CCTA and evaluate the association of cardiac and non-cardiac imaging with laboratory markers and clinical data including outcome.

DETAILED DESCRIPTION:
In this study the investigators retrospectively and prospectively collect information from enrolled subjects through a period of a total of 10 years to evaluate multidimensional associations between phenotypic manifestations of cardiovascular disease via CCTA and cardiac and non-cardiac imaging, serum biomarkers, demographic and clinical information, clinical presentation (cross-sectional), therapy changes (time-varying) and their ability to predict mortality and MACE (major adverse cardiac event ) (longitudinal) in patients clinically indicated for CCTA.

The aim is to establish a comprehensive cross-sectional, time-varying and longitudinal data collection for individuals undergoing clinically-indicated CCTA to date in order to apply novel multiparametric approaches to determine cardiovascular significance to clinically-important patient-centered events. For data collection this registry will follow a standard CRF (case report form) structure, so to enable the merging of this data-set with other international registries, which might contribute in overcoming some gaps of knowledge from previous CCTA studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult individual >18 years
* Undergoing clinically indicated CCTA
* Signed informed consent or waiver

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry foreseen a prospective cohort composed by patients undergoing clinically indicated CCTA and by a retrospective population of patients that have undergone CCTA 1st June 2017 to 31st December 2020. The principal investigator confirms that no patient's personal health data will be collected if a written or documented oral refusal exist.
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2031-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death. | 10 years
  The primary endpoint is the time to first occurrence of death from all-causes.

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 10 years
  The secondary composite endpoint is major adverse cardiac events (MACE), which is defined by the occurrence of any of the following events:
  1. All-cause death
  2. Myocardial infarction
  3. Unstable angina-related hospitalization
  4. Late coronary revascularization (≥90 days)
Other outcome | 10 years
  Occurrence of any of the following events:
  1. Cerebrovascular accident
  2. Valvular intervention
  3. Congestive heart failure-related hospitalization
  4. Cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, MD, PhD, Principal Investigator — Department of Cardiology, University Hospital Bern,
Locations (1):
- Department of Cardiology, University Hospital Bern, Inselspital, Bern, Bern, Switzerland